CLINICAL TRIAL: NCT03399149
Title: Systematic Evaluation by an Intensivist of Hematological Malignancy Patients Presenting With Acute Respiratory or Hemodynamic Failure: Impact on Prognosis: A Monocentric Observational Before-after Study
Brief Title: Systematic Evaluation by an Intensivist of Hematological Malignancy Patients Presenting With Acute Respiratory or Hemodynamic Failure
Acronym: CAREHEMA
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: CARE HEMA (38RC16.238); 2017-A00411-52 (Other: ID RCB)
Record Dates: First submitted 2017-12-01; First posted 2018-01-16 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-06

CONDITIONS: Respiratory Insufficiency; Hematologic Malignancy
Keywords: Respiratory Insufficiency; Hematologic Malignancy; Intensive Care Unit
MeSH Terms: conditions — Respiratory Insufficiency; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- "Before phase": Retrospective study of ICU admissions of hematology patients for respiratory and hemodynamic reasons Time period: January 2012 to March 2017
- "After Phase": Systematic evaluation by an intensivist: Corresponding to the period after the implementation of a systematic intensivist evaluation Daily screening of systolic blood pressure, oxygen saturation and oxygen requirements of all patients hospitalized in hematology wards. Systematic evaluation of any patient presenting the inclusion criteria by an intensivist and collegial care planning.
  Time period: From March 2017 to end of study
  Interventions: Other: Systematic evaluation by an intensivist

INTERVENTIONS:
Other: Systematic evaluation by an intensivist — implementation of a standardized procedure for patient care in ICU
  Groups: "After Phase": Systematic evaluation by an intensivist

SUMMARY:
Over the last two decades, the number of patients with hematological malignancies (HMs) admitted to the ICU increased and their mortality has dropped sharply. Patients with HMs increasingly require admission to the intensive care unit (ICU) for life-threatening events related to the malignancy and/or treatments, with immunosuppression being a major contributor. Whether the increase in ICU admissions is related to increased referrals by hematologists and/or to increased admissions by intensivists is unknown. The criteria used for ICU referral and admission decisions have not been extensively evaluated. Finally, the links between admission policies and treatment-limitation decisions are unclear, but ICUs with broad admission policies may change the treatment goals based on the response to several days of full-code management.

The aim of this study is to evaluate the impact of a systematic evaluation by an intensivist of HMs patients presenting with acute respiratory and/or hemodynamic failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in a hematology unit
* Patients presenting with criteria for critical respiratory and/or hemodynamic condition and worsening during the next 4 hours

  1. Respiratory : oxygen saturation <90 % and/or O2 >3l/min, with either a worsening of saturation or increased oxygen needs within 4h
  2. Hemodynamic : systolic blood pressure < 90 mmHg and remaining < 90 mmHg within 4h despite ≥ 1l of crystalloid administration, or becoming < 80 mmHg no matter the quantity of fluid (even if no fluid administration).

Exclusion Criteria:

* therapeutic limitations decided hematological investigators (moribund patients, uncontrolled allogenic graft,...)
* Do-not-reanimate directives
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with haematological malignacies, presenting acute respiratory and/or hemodynamic failure
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
delta Sepsis-related Organ Failure Assessment (SOFA) score | up to 72 hours
  difference between the Sepsis-related Organ Failure Assessment score between 48h and 72h after ICU admission and the SOFA score during the first 24h.
  SOFA score ranges from 0 to 20 delta SOFA= SOFA day 3 - SOFA day1

SECONDARY OUTCOMES:
survival status after one year | one year after ICU admission
  survival status (alive/dead) at one year after ICU admission
survival status at the end of the ICU stage | up to Day 45
  survival status (alive/dead) at the end of the ICU stage
survival status at the end of the hospitalization | up to Day 120
  survival status (alive/dead) at the end of the hospitalization
ICU admission | up to 72h
  Delay between the start of critical care illness and ICU admission Delay is measured in minutes
Invasive mechanical ventilation | up to Day 45
  Number of days with mechanical ventilation
Non-invasive ventilation | up to Day 45
  Number of days with non-invasive ventilation
Vasopressive support | up to Day 45
  Number of days with vasopressive support
renal replacement therapy | up to Day 45
  Number of days with renal replacement therapy
hematological disease evolution | up to one year
  status of hematological primary disease at death or after one year of evolution if the patient is still alive. Possible status of hematology disease : complete remission, partial remission, stability, relapsed/refractory.
Life quality for patients | up to one year
  EQ5-D assessment of patients' quality of life one year after Intensive care unit admission

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Terzi, Principal Investigator — CHU Grenoble Alpes
Locations (2):
- France (2):
  - Hematologic unit - Hospital Grenoble Alpes, Grenoble
  - Intensive Care Unit - Hospital Grenoble-Alpes, Grenoble